# **Cover Page for SAP**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT04083781 |
| Sponsor trial ID: | NN7415-4311 |
| Official title of study: | Efficacy and safety of concizumab prophylaxis in patients with haemophilia A or B with inhibitors |
| Document date* | 27-Jul-2022 |

<sup>\*</sup>Document date refers to the date on which the document was most recently updated.

Statistical Analysis Plan W56 Trial ID: NN7415-4311 UTN: U1111-1225-9670 EudraCT No.: 2018-004889-34 
 Date:
 21 July 2022
 Novo Nordisk

 Version:
 2.0

 Status:
 Final

 Page:

## NN7415-4311

# Statistical Analysis Plan Week 56 cut-off

Redacted protocol Includes redaction of personal identifiable information only.

, Statistician Biostatistics, Biopharm 1

Statistical Analysis Plan W56 Trial ID: NN7415-4311 UTN: U1111-1225-9670 EudraCT No.: 2018-004889-34 Date: Version: Status: Page:

2.0 Final 2 of 26

# **Table of contents**

| | | | Page |
|---|---|---|---|
| Га | ble of | contents | 2 |
| Га | ble of | tables | 3 |
| Ve | rsion l | history | 4 |
| 1 | Intro | oduction | 5 |
| | 1.1 | Objectives and endpoints | |
| | 1.2 | Trial design | |
| 2 | Stati | stical hypotheses | 8 |
| 3 | Samj | ple size determination | 9 |
| 1 | Anal | ysis sets | 10 |
| 5 | Stati | stical analyses | 12 |
| | 5.1 | General considerations. | |
| | 5.2 | Subject disposition | 13 |
| | 5.3 | Primary endpoint analysis | 13 |
| | 5.4 | Secondary endpoint analysis | 13 |
| | 5.5 | | |
| | | 5.5.1 Bleed-related assessments | |
| | | 5.5.2 Pharmacokinetic and pharmacodynamic assessments | |
| | 5.6 | Exploratory safety analyses | |
| | | 5.6.1 Extent of exposure | |
| | | 5.6.2 Adverse events | |
| | | 5.6.3 Additional safety assessments | |
| | 5.7 | Subgroup analyses | |
| | 5.8 | Interim analyses | |
| | | 5.8.1 Data monitoring committee | 16 |
| 6 | Supp | oorting documentation | 17 |
| | 6.1 | Appendix 1: List of abbreviations | |
| | 6.2 | Appendix 2: Definition of exploratory efficacy/safety endpoints and assessments | 18 |
| 7 | Dofo | renees Error! Poolsmark no | t defined |

 Statistical Analysis Plan W56
 Date:
 21 July 2022
 Novo Nordisk

 Trial ID: NN7415-4311
 Version:
 2.0

 UTN: U1111-1225-9670
 Status:
 Final

 EudraCT No.: 2018-004889-34
 Page:

# **Table of tables**

| | | Page |
|---|---|---|
| Table 1 | Analysis sets used for analyses and/or presentations of endpoints/assessments | 12 |

 Statistical Analysis Plan W56
 Date:
 21 July 2022
 Novo Nordisk

 Trial ID: NN7415-4311
 Version:
 2.0

 UTN: U1111-1225-9670
 Status:
 Final

 EudraCT No.: 2018-004889-34
 Page:

# **Version history**

This Statistical Analysis Plan (SAP) describes the data evaluation planned for the 56 weeks cut-off as mentioned in the NN7415-4311 trial protocol version 7.0 (dated 18-Jun-2021).

| SAP<br>Version | Approval<br>Date | Change | Rationale |
|---|---|---|---|
| 1 | 18-Dec-2019 | Not Applicable | Original version |
| 2 | 27-Jul-2022 | Updated Description for<br>Defined Analysis Data Set<br>"On-treatment" in section 4 | Second bullet of the "Ontreatment" analysis data set in section 4, was not updated when updating SAP from primary analysis cut-off to 56 weeks cut-off. Wording in second bullet has now been changed from "The last direct subject-site contact, at or prior to the <i>primary analysis</i> cut-off" to "The last direct subject-site contact, at or prior to the <i>56 weeks</i> cut-off". |

 Statistical Analysis Plan W56
 Date:
 21 July 2022
 Novo Nordisk

 Trial ID: NN7415-4311
 Version:
 2.0

 UTN: U1111-1225-9670
 Status:
 Final

 EudraCT No.: 2018-004889-34
 Page:

#### 1 Introduction

This SAP describes descriptive analyses for the endpoints/assessments related to bleeding episodes, safety and PK/PD for the evaluation made at the 56-week cut-off of trial NN7415-4311. The 56-week cut-off is defined as when all patients in arms 2, 3 and 4 have completed visit 13a (or permanently discontinued treatment). For a description of the analyses planned for the main part of the trial please refer to the SAP for the primary analysis cut-off.

All confirmatory conclusions for this trial are based on the analyses done at the primary analysis cut-off. No further confirmatory conclusions can be made based on the descriptive analyses described in this SAP.

Additional details on the derivation and calculation based on the measurements collected in this trial will be described in the analysis data reviewer's guide (ADRG). In addition, specifications of tables, figures and listings (TFL) are described in the mock TLFs.

Note, in this document 'bleeds' refer to 'bleeding episodes'.

 Statistical Analysis Plan W56
 Date:
 21 July 2022
 Novo Nordisk

 Trial ID: NN7415-4311
 Version:
 2.0

 UTN: U1111-1225-9670
 Status:
 Final

 EudraCT No.: 2018-004889-34
 Page:

#### 1.1 Objectives and endpoints

No specific objectives are defined to specifically relate to the 56 weeks cut off. For the objectives related to PACO, please refer to the protocol.

All the details of the endpoints, assessments and timeframes for the week 56 cut-off are explained in the appendix 2.

 Statistical Analysis Plan W56
 Date:
 21 July 2022
 Novo Nordisk

 Trial ID: NN7415-4311
 Version:
 2.0

 UTN: U1111-1225-9670
 Status:
 Final

 EudraCT No.: 2018-004889-34
 Page:

#### 1.2 Trial design

The following is a brief sum up of the most important parts of the trial design. For further details refer to the trial protocol version 7.

- This is a prospective, multicentre, open label clinical trial with four arms with the aims to evaluate the effect and safety of daily concizumab prophylaxis administered s.c. in subjects with HAwI and HBwI. The four arms of the trial consist of:
  - o Arms 1 and 2 consist of subjects previously treated on demand who are randomised to
    - Arm 1: On-demand administration
    - Arm 2: Concizumab PPX treatment
  - Arms 3 and 4 are allocated to receive concizumab PPX treatment and consist of subjects who are
    - Arm 3: Transferred from trial 4310
    - Arm 4: Previously treated on PPX or on demand
- In the second quarter of 2020, the protocol was amended (protocol version 3.0) to incorporate measures to mitigate the risk of thromboembolic events. These measures include the handling of factor treatment for BTB and changes to the dosing regimen. As a result of these changes and the pause in the treatment while the protocol was to be amended, all statistical analyses were reconsidered and adjusted accordingly.
- The primary analysis is made when all subjects in arm 1 have completed visit 9/9a (or withdrawn) and all subjects in arm 2 have completed visit 10a (or withdrawn).
- After the main part of the trial, all patients have offered to continue in the extension part of the trial and receive treatment with concizumab for up to an additional 128 weeks (arms 2-4) or 136 weeks (arm 1)
- After 56 weeks of treatment in arms 2, 3 and 4, an additional evaluation will be made assessing bleed-related endpoints and safety for concizumab. This SAP describes in more detail the descriptive analyses that are relevant for this cut-off.
- After the last patient has been randomised, any patient that due to the COVID-19 pandemic is
  prevented from restarting the new dosing regimen will no longer be used to determine the
  primary analysis cut-off and the 56-week cut-off.

 Statistical Analysis Plan W56
 Date:
 21 July 2022
 Novo Nordisk

 Trial ID: NN7415-4311
 Version:
 2.0

 UTN: U1111-1225-9670
 Status:
 Final

 EudraCT No.: 2018-004889-34
 Page:

# 2 Statistical hypotheses

For the analyses related to the week 56 cut-off no statistical hypotheses are tested.

#### **Multiplicity Adjustment**

No adjustment for multiplicity is needed since no statistical hypotheses are tested.

 Statistical Analysis Plan W56
 Date:
 21 July 2022
 Novo Nordisk

 Trial ID: NN7415-4311
 Version:
 2.0

 UTN: U1111-1225-9670
 Status:
 Final

 EudraCT No.: 2018-004889-34
 Page:

# 3 Sample size determination

The sample size considerations are described in detail in section 10.1 of the protocol version 7.

| Statistical Analysis Plan W56 | Date: | 21 July 2022 Novo Nordisk |
|-------------------------------|----------|---------------------------|
| Trial ID: NN7415-4311 | Version: | 2.0 |
| UTN: U1111-1225-9670 | Status: | Final |
| EudraCT No.: 2018-004889-34 | Page: | 10 of 26 |

#### **Analysis sets** 4

For the purposes of analysis, the following analysis sets are defined for the week 56 cut-off.

| Subject Analysis<br>Set | Description |
|---|---|
| Full Analysis Set (FAS) | All subjects randomised to concizumab PPX or on-demand treatment or allocated to arms 3 or 4. Subjects from arms 1 and 2 will contribute to the evaluation 'as randomised'. |
| Safety Analysis Set (SAS) | All subjects exposed to concizumab PPX or randomised to on-demand treatment. All subjects will contribute to the evaluation 'as treated'. |

| Defined Analysis<br>Data Sets | Description |
|---|---|
| On-treatment | The time period where subjects are considered to be affected by on-<br>demand treatment or concizumab treatment. |
| | For safety endpoints/assessments relating to events (number of thromboembolic events, number of hypersensitivity type reactions, number of injection site reactions, number of patients with antibodies to concizumab, number of adverse events) the 'on-treatment' analysis data set is defined as follows. |
| | For subjects in <b>arm 1 during on-demand treatment</b> , the period begins on the date of randomisation (as registered in IWRS) and ends at the first occurrence of: |
| | <ol> <li>Time of permanently ending on-demand administration and initiation of any PPX regimen</li> <li>The last direct subject-site contact, at or prior to the 56 weeks cut-off</li> <li>Withdrawal date for subjects who withdraw informed consent</li> <li>The last subject-investigator/site contact as defined by investigator for subjects who are completely lost to follow up</li> <li>Date of death for subjects</li> </ol> |
| | For subjects in <b>arm 1 during concizumab PPX treatment</b> , the period begins at the time of initiation of concizumab PPX treatment and ends at the first occurrence of: |
| | <ul> <li>6. Date of last dose of concizumab + 7 weeks</li> <li>7. Items 2., 3., 4. or 5. above</li> </ul> |
| | For subjects in arms 2-4 that start on the new concizumab dosing regimen and who have not been exposed to the initial dosing regimen, the period begins at the time of start of the new concizumab PPX regimen. |

Trial ID: NN7415-4311 UTN: U1111-1225-9670 EudraCT No.: 2018-004889-34

| ı | i age. | 11 01 20 |
|---|---|---|
| For subjects in arms 2-4 that a | are only exposed | to the initial |
| concizumab dosing regimen, | the period begins | at the time of start of |
| the initial concizumab PPX reg | gimen. | |

Status:

Final


For subjects in arms 2-4 that start on the new concizumab dosing regimen and who have been exposed to the initial dosing regimen, the period consists of two periods with a pause in between. The first period begins at the time of start of the initial concizumab PPX regimen and ends 7 weeks after the treatment was paused while the second period begins at the time of start of the new concizumab PPX regimen.

For all cases of arms 2-4 above the periods end at the first occurrence of:

• Items 2., 3., 4., 5. or 6. above

# On-treatment without data on initial regimen

The time period where subjects are considered to be affected by ondemand treatment or treatment with the new concizumab dosing regimen.

The analysis data set is defined similarly as the 'on-treatment' analysis data set with the exception:

• Observation time during the initial concizumab PPX regimen is excluded

# On-treatment without ancillary therapy<sup>a</sup> excl. data on initial regimen for subjects exposed to both regimens

The time period where subjects are treated by either the new concizumab dosing regimen or the initial concizumab dosing regimen (only included if not exposed to the new concizumab dosing regimen) or are treated by on-demand treatment and additionally have not used factor-containing products not related to treatment of a bleed during any of the cases.

The analysis data set is defined similarly as the 'on-treatment' analysis data set with the exception:

- Periods where factor containing products not related to treatment of a bleed have been used are excluded
- For subjects in arms 2-4 that start on the new concizumab dosing regimen and who have been exposed to the initial dosing regimen, the data on the initial concizumab PPX regimen are excluded

<sup>&</sup>lt;sup>a</sup> Ancillary therapy is defined as use of factor-containing products not related to treatment of a bleed.

Statistical Analysis Plan W56 Date: 21 July 2022 Novo Nordisk Version: Final


UTN: U1111-1225-9670 Status: EudraCT No.: 2018-004889-34 Page:

#### Statistical analyses 5

Trial ID: NN7415-4311

#### 5.1 **General considerations**

This SAP will address the details of the descriptive statistics implemented on all arms (1, 2, 3 and 4) at the 56-week cut-off of trial NN7415-4311. The 56-week cut-off is defined as when all patients in arms 2, 3 and 4 have completed visit 13a (or permanently discontinued treatment). After the last patient has been randomised, any patient that due to the COVID-19 pandemic is prevented from restarting the new dosing regimen will no longer be used to determine the 56-week cut-off.

Unless specified otherwise, the endpoints/assessments will be presented using the analysis sets as displayed in Table 1.

Table 1 Analysis sets used for analyses and/or presentations of endpoints/assessments

| Endpoint/assessment categories <sup>a</sup> | Subject<br>Analysis Set | Analysis Data Sets |
|---|---|---|
| Bleeding episodes | FAS | On-treatment without ancillary therapy excl. data on initial regimen for subjects exposed to both regimens |
| PK, PD and safety not relating to events | SAS | On-treatment without data on initial regimen |
| Safety relating to events <sup>b</sup> | SAS | On-treatment and On-treatment without data on initial regimen |

<sup>&</sup>lt;sup>a</sup>Which endpoints/assessments that belong under each category can be found in section 9 of the protocol version 7. <sup>b</sup>This specifically refers to: number of thromboembolic events, number of hypersensitivity type reactions, number of injection site reactions, number of patients with antibodies to concizumab, and number of adverse events.

For arms 2-4 the target joints registered at baseline will be used for the assessment done at week 56. For arm 1 the target joint evaluation done at visit V9a will be used for assessment at week 56.

Continuous endpoints/assessments will be presented using descriptive statistics which will include min, max, mean, SD, median, and quartiles. For PK endpoints/assessments, the descriptive statistics will also include geometric mean and geometric CV. Event data (including AEs) will be summarised including number of subjects with an event/episode, percentage of subjects with an event/episode, number of events/episodes and rate of events/episodes. Categorical assessments will be summarised by number and percent of subjects in each category. Presentations of results will be by arm and visit (when applicable) and when relevant arm 1 will be split into two parts with ondemand treatment and concizumab treatment.

Baseline for the assessments done at week 56 is defined as the latest non-missing measurement recorded before the time of the first administration of concizumab with the new dosing regimen (arms 2-4 and arm 1 after receiving concizumab) or recorded before randomisation to the ondemand administration (arm 1). If this measurement is missing for arms 2-4 or a subject from arms 2-4 chooses not to restart on concizumab, then the baseline obtained prior to the initial dosing regimen will be used (if available). If the V9a measurement is missing for arm 1 concizumab part,

| Statistical Analysis Plan W56 | Date: | 21 July 2022 | Novo Nordisk |
|-------------------------------|----------|--------------|--------------|
| Trial ID: NN7415-4311 | Version: | 2.0 | |
| UTN: U1111-1225-9670 | Status: | Final | |
| EudraCT No.: 2018-004889-34 | Page: | 13 of 26 | |

the latest measurement recorded prior to V9a will be used as a concizumab baseline for arm 1 subjects.

As described in the protocol, if a patient withdraws from trial prior to visit 9/9a/10a (last treatment visit in the main part of the trial), the investigator should ask the patient if he is willing, as soon as possible, to have assessment performed according to visit 9/9a/10a. If the patient withdraws from trial after visit 9a/10a, he should have assessment performed according to visit 26a (last treatment visit in the extension part of the trial). Any values obtained because of this are in scope for being reallocated to a (planned) scheduled visit. Only the value(s) that fulfil the below reallocation rules can be used in summaries and the analyses. The value(s) will be reallocated to a (planned) scheduled visit if the following apply:

- The visit falls within an extended visit window of +/- 7 days of the (planned) scheduled visit.
- The same parameter was planned for assessment but was not assessed at the scheduled visit.
- The scheduled visit is neither a screening visit (visit 1/1a), a randomisation visit (visit 2/2a) or a V9/V9a (only relevant if the patient withdraws from the trial after V9a/10a).

In terms of bleed related endpoints, the bleed rate is defined as the number of bleeds over the respective observation periods. Multiple bleeding locations at the same time point will be counted as one bleeding episode. As a general rule, a treated bleed is defined as any bleed where the use of a factor-containing product is reported between the start and stop time of a bleed. Further, the endpoints will not include re-bleeds. A re-bleed is defined as a bleeding episode (worsening of bleeding site conditions e.g. swelling, pain) starting within 72 hours after stopping treatment of a previous treated bleeding episode (or re-bleed) at the same anatomical location. Note that there can be more than one re-bleed related to the same bleed. If a bleeding episode occurs in the same location more than 72 hours after stopping treatment of a previous bleeding episode (or re-bleed) in the same location, the bleed is defined as a new bleeding episode.

Pharmacokinetic concentration values below lower limit of quantification (LLOQ) is handled as described below:

| Timing of values below LLOQ | Imputation | Use of imputed |
|---|---|---|
| | | values |
| Values below LLOQ obtained before time of the first administration with the initial dosing regimen and with the new dosing regimen | Set to 0 (zero) | Plots and derivation of AUC |
| All other values below LLOQ | Set to LLOQ/2 | Plots and derivation of AUC |

#### 5.2 Subject disposition

See mock TFLs.

#### 5.3 Primary endpoint analysis

Refer to SAP for PACO.

#### 5.4 Secondary endpoint analysis

Refer to SAP for PACO.

| Statistical Analysis Plan W56 | Date: | 21 July 2022 | Novo Nordisk |
|-------------------------------|----------|--------------|--------------|
| Trial ID: NN7415-4311 | Version: | 2.0 | |
| UTN: U1111-1225-9670 | Status: | Final | |
| EudraCT No.: 2018-004889-34 | Page: | 14 of 26 | |

#### 5.5 Exploratory efficacy endpoints analysis

#### 5.5.1 Bleed-related assessments

The assessments related to bleeding episodes are defined in section 6.2.

The definition of bleeding rate, treated bleeds and re-bleeds are defined in the section <u>5.1</u> of this document and in section 10.3 of protocol version 7. The definition of a target joint is given in the protocol section 9.1.4.

ABR will be calculated at an individual basis as

$$ABR = \left(\frac{\text{Number of treated spontaneous or traumatic bleeds}}{\text{Number of days in the analysis data set}}\right) x 365.25$$

The continuous/categorical assessments will be presented using descriptive statistics as described in section <u>5.1</u>. The descriptive statistics for the bleed related assessments up until week 56 will be presented by treatment arms and 'Total concizumab'. Furthermore, it will be presented by haemophilia types (HAwI, HBwI).

The evaluation of bleeding episodes at target joints up until 56 weeks will be done between treatment arms and as 'Total concizumab'.

These descriptive statistics tables will enumerate results for treated bleeds, zero treated bleeds, cause of bleeds (Spontaneous, Traumatic, Surgical), anatomical location of bleeds (Target joints, Joints, Muscular, Skin, Gastrointestinal, Mouth-gums-nose, Urinary system, Central nervous system, Other), classification of bleeds (Mild/moderate, Severe) and location of severe bleeds (Target joints, Joints, Muscular, Skin, Gastrointestinal, Mouth-gums-nose, Urinary system, Central nervous system, Other). The analysis data set use for these descriptive statistics are mentioned in section 5.1 of this document.

#### 5.5.2 Pharmacokinetic and pharmacodynamic assessments

The assessments related to PK and PD are defined in section 6.2.

Concizumab concentrations collected during the trial will be used to derive the pharmacokinetic endpoints and assessments based on non-compartmental methods.

All PK and PD endpoints and assessments are continuous and will be presented using the descriptive statistics and analysis sets as described under section 5.1.

 Statistical Analysis Plan W56
 Date:
 21 July 2022
 Novo Nordisk

 Trial ID: NN7415-4311
 Version:
 2.0

 UTN: U1111-1225-9670
 Status:
 Final

Page:


UTN: U1111-1225-9670 EudraCT No.: 2018-004889-34

#### 5.6 Exploratory safety analyses

#### 5.6.1 Extent of exposure

A summary showing subjects that escalate, deescalate, or remain on the 0.20 mg/kg/day dose will be presented by arm.

The length of the periods constituting the analysis data sets and the number of doses taken will be presented descriptively. The output will differentiate between before the pause, after the pause and in total.

#### **5.6.2** Adverse events

All exploratory safety endpoints are defined in section 6.2.

All adverse events will be coded using the current version of MedDRA. Hypersensitivity reactions, medication errors and injection site reactions are categorised in the CRF as AEs requiring additional data collection. Additional information on these events will be collected using separate forms. Further, a MedDRA search will also be used to define these events. Thromboembolic events are defined and categorised as AESIs.

Adverse events will be evaluated using descriptive statistics based on the analysis data sets as described in section <u>5.1</u>. These descriptive statistics tables will also be presented by treatment arms and 'Total concizumab'.

Furthermore, for the on-treatment analysis data set the outputs on adverse events will also include information on

- System organ class
- Severity (mild/moderate/severe), seriousness (serious/non-serious) and relation to treatment (possibly/probably/unlikely)
- Adverse events leading to drug discontinuation
- Most frequent adverse events (occurring in more or equal to 5% of subjects)
- Deaths
- Medication errors

The outputs may differentiate between the initial part of the trial and the part after the restart of the trial if deemed relevant.

#### 5.6.3 Additional safety assessments

Assessments in relation to planned safety laboratory measurement, body measurements, vital signs and physical examinations are defined in section  $\underline{6.2}$ . The assessments will be presented using descriptive statistics as described in section  $\underline{5.1}$ . Number of patients with a positive antibody test will be presented as described in section  $\underline{5.1}$  and furthermore a list of all positive antibodies recorded during the trial will be presented.

| Statistical Analysis Plan W56 | Date: | 21 July 2022 Novo Nordisk |
|-------------------------------|----------|-----------------------------|
| Trial ID: NN7415-4311 | Version: | 2.0 |
| UTN: U1111-1225-9670 | Status: | Final |
| EudraCT No.: 2018-004889-34 | Page: | 16 of 26 |

#### 5.7 Subgroup analyses

Descriptive statistics by subgroups are specified for haemophilia types (HAwI or HBwI) above in each of the sections concerning the specific assessments, such as bleed related endpoints.

#### 5.8 Interim analyses

No formal interim analyses are planned.

Several evaluations are to be made during the conduct of the trial:

- at the primary analysis cut-off
- after 56 weeks
- at the end of the extension part

After the initial evaluation at the primary analysis cut-off no further confirmatory conclusions can be made.

#### **5.8.1** Data monitoring committee

A Data Monitoring Committee (DMC) is established to review and evaluate accumulating data from the trial in order to protect the safety of the subjects.

The DMC members are not having direct contact with any Novo Nordisk staff involved with the trial except for Novo Nordisk global safety. Details in relation to DMC can be seen in Appendix 4 of the protocol version 7.

Statistical Analysis Plan W56 Trial ID: NN7415-4311 UTN: U1111-1225-9670 EudraCT No.: 2018-004889-34 

 Date:
 21 July 2022

 Version:
 2.0

 Status:
 Final

 Page:

Novo Nordisk

## 6 Supporting documentation

#### 6.1 Appendix 1: List of abbreviations

ABR Annual Bleeding Rate

ADRG Analysis Data Reviewer's Guide

AE Adverse event

AESI Adverse event of special interest

AUC Area under the curve

DMC Data monitoring committee

FAS Full analysis set

HAwI Haemophilia A with inhibitors
HBwI Haemophilia B with inhibitors
IWRS interactive web response system
LLoQ Lower limit of quantification

MedDRA Medical dictionary for regulatory activities

PACO Primary analysis cut-off

PD Pharmacodynamic
PK Pharmacokinetic
PPX Prophylaxis

SAP Statistical Analysis Plan

SAS Safety analysis set

TFL tables, figures and listings

TFPI Tissue factor pathway inhibitor

Statistical Analysis Plan W56 Trial ID: NN7415-4311

UTN: U1111-1225-9670 EudraCT No.: 2018-004889-34

Date: Version:

21 July 2022 | Status: 2.0 | Page:

Final Novo Nordisk

#### Appendix 2: Definition of exploratory efficacy/safety endpoints and assessments **6.2**

| Type | Title | Time frame | Unit | Details | Section |
|---|---|---|---|---|---|
| Assessment | Number of<br>treated<br>spontaneous<br>and traumatic<br>bleeding<br>episodes | On demand (arm 1) • From randomisation (week 0) up until start of concizumab treatment (at least 24 weeks) | Count | Week 56 cut-off is when all patients from arm 2-4 have completed visit 13a assessments or permanently discontinued treatment. Concizumab (arm 1) data available up until week 56 cut-off will be presented. | 5.5.1 |
| | | Concizumab (arm 1) • From start of the new concizumab dosing regimen up until week 56 cut-off Concizumab (arms 2-4) | | | |
| | | • From start of the new concizumab dosing regimen (week 0) up until week 56 cut-off | | | |
| Assessment | Number of<br>treated<br>spontaneous<br>bleeding<br>episodes | On demand (arm 1) • From randomisation (week 0) up until start of concizumab treatment (at least 24 weeks) | Count | Week 56 cut-off is when all patients from arm 2-4 have completed visit 13a assessments or permanently discontinued treatment. Concizumab (arm 1) data available up until week 56 cut-off will be presented. | 5.5.1 |
| | | <ul> <li>Concizumab (arm 1)</li> <li>From start of the new concizumab dosing regimen up until week 56 cut-off</li> </ul> | | | |

| Statistical Analys<br>Trial ID: NN741 | | UTN: U1111-1225-9670<br>EudraCT No.: 2018-004889-34 | Date:<br>Version: | 21 July 2022<br>2.0 | | inal<br>f 26 | Novo Nordisk |
|---|---|---|---|---|---|---|---|
| | | Concizumab (arms 2-4) • From start of the new concizumab dosing regimen (week 0) up until week 56 cut-off | | | | | |
| Assessment | Number of treated spontaneous and traumatic joint bleeds | On demand (arm 1) • From randomisation (week 0) up until start of concizumab treatment (at least 24 weeks) Concizumab (arm 1) • From start of the new concizumab dosing regimen up until week 56 cut-off Concizumab (arms 2-4) • From start of the new concizumab dosing regimen (week 0) up until week 56 cut-off | Count | 2-4 have complete permanently disco | s when all patients from armed visit 13a assessments or ontinued treatment. 1) data available up untilizill be presented. | m | 5.5.1 |
| Assessment | Number of<br>treated<br>spontaneous<br>and traumatic<br>target joint<br>bleeds | On demand (arm 1) • From randomisation (week 0) up until start of concizumab treatment (at least 24 weeks) Concizumab (arm 1) | Count | 2-4 have complete permanently disco | s when all patients from armed visit 13a assessments or ontinued treatment. 1) data available up until vill be presented. | n | 5.5.1 |

| Statistical Analys<br>Trial ID: NN741 | | UTN: U1111-1225-9670<br>EudraCT No.: 2018-004889-34 | Date:<br>Version: | 21 July 2022<br>2.0 | Status: Final Page: 20 of 26 | |
|---|---|---|---|---|---|---|
| | | From start of the new concizumab dosing regimen up until week 56 cut-off | | | | |
| | | <ul> <li>Concizumab (arms 2-4)</li> <li>From start of the new concizumab dosing regimen (week 0) up until week 56 cut-off</li> </ul> | | | | |
| Assessment | The number of all spontaneous and traumatic bleeds (treated and untreated) | On demand (arm 1) From randomisation (week 0) up until start of concizumab treatment (at least 24 weeks) Concizumab (arm 1) From start of the new concizumab dosing regimen up until week 56 cut-off Concizumab (arms 2-4) From start of the new concizumab dosing regimen (week 0) up until week 56 cut-off | Count | 2-4 have complete permanently disco | s when all patients from arm ed visit 13a assessments or ontinued treatment. 1) data available up until vill be presented. | 5.5.1 |
| Assessment | Pre-dose<br>concizumab<br>plasma<br>concentration | Concizumab (arms 2-4) • From start of the new concizumab dosing | ng/mL | | dose assessments from start umab dosing regimen (week 66. | 5.5.2 |

| Statistical Analys<br>Trial ID: NN741 | | UTN: U1111-1225-9670<br>EudraCT No.: 2018-004889-34 | Date:<br>Version: | 21 July 2022<br>2.0 | Status:<br>Page: | Final<br>21 of 26 | Novo Nordisk |
|---|---|---|---|---|---|---|---|
| | | regimen (week 0) up<br>until week 56 cut-off | | | | | |
| Assessment | Thrombin peak | At visits where thrombin generation assessments are planned to be measured in the trial up to 56 weeks | nmol/L | 56. | e assessments up until<br>new concizumab dosir<br>up until week 56. | | <u>5.5.2</u> |
| Assessment | Free TFPI concentration | At visits where free TFPI assessments are planned to be measured in the trial up to 56 weeks | ng/mL | | | | 5.5.2 |
| Assessment | Endogenous<br>thrombin<br>potential (ETP) | At visits where thrombin generation assessments are planned to be measured in the trial up to 56 weeks | nmol/L*min | | | | 5.5.2 |
| Assessment | Endogenous<br>thrombin<br>Potential ratio | At visits where thrombin generation assessments are planned to be measured in the trial up to 56 weeks | Ratio | | | | 5.5.2 |
| Assessment | Velocity index | At visits where thrombin generation assessments are planned to be measured in the trial up to 56 weeks | nmol/L*min | | | | 5.5.2 |
| Assessment | Thrombin lag time | At visits where thrombin generation assessments are planned to be measured in the trial up to 56 weeks | min | | | | 5.5.2 |

| Statistical Analys<br>Trial ID: NN741 | | UTN: U1111-1225-9670<br>EudraCT No.: 2018-004889-34 | Date:<br>Version: | 21 July 2022<br>2.0 | Status: Fina Page: 22 of 20 | |
|---|---|---|---|---|---|---|
| Assessment | Time to thrombin peak | At visits where thrombin generation assessments are planned to be measured in the trial up to 56 weeks | min | | | 5.5.2 |
| Assessment | Number of adverse events | On demand (arm 1) • From randomisation | Count | | s when all patients from arm ed visit 13a assessments or | 5.6.2 |
| Assessment | Number of thromboembolic events | to on demand<br>treatment up until start<br>of concizumab | Count | | ontinued treatment. 1) data available up until | 5.6.2 |
| Assessment | Number of hypersensitivity type reactions | treatment Concizumab (arm 1) | Count | week 56 cut-off w | vill be presented. | 5.6.2 |
| Assessment | Number of injection site reactions | <ul> <li>From start of the new concizumab dosing regimen up until week 56 cut-off</li> <li>Concizumab (arms 2-4)</li> <li>Before the pause: <ul> <li>From start of concizumab treatment (week 0) up until 7 weeks after the treatment pause</li> </ul> </li> <li>as well as</li> <li>After the pause: From start of the new concizumab treatment (week 0) up until week 56 cut-off</li> </ul> | Count | | | 5.6.2 |

| Statistical Analys<br>Trial ID: NN741 | | UTN: U1111-1225-9670<br>EudraCT No.: 2018-004889-34 | Date:<br>Version: | 21 July 2022 Status:<br>2.0 Page: | Final 23 of 26 | Novo Nordisk |
|---|---|---|---|---|---|---|
| Assessment | Number of patients with antibodies to concizumab | <ul> <li>Concizumab (arms 2-4)</li> <li>From start of the new concizumab dosing regimen (week 0) up until week 56 cut-off</li> </ul> | Count | Week 56 cut-off is when all patients for 2-4 have completed visit 13a assessmit permanently discontinued treatment. | | 5.6.3 |
| Assessment | Change in<br><safety<br>laboratory<br/>parameter&gt;</safety<br> | <ul> <li>On demand (arm 1)</li> <li>From randomisation (week 0) up until start of concizumab treatment (at least 24 weeks)</li> <li>Concizumab (arm 1)</li> <li>From start of the new concizumab dosing regimen up until week 56 cut-off</li> <li>Concizumab (arms 2-4)</li> <li>From start of the new concizumab dosing regimen (week 0) up until week 56 cut-off</li> <li>From start of treatment (week 0) to every visit where the <safety laboratory="" parameter=""> is planned to be measured up until V13a (week 56)</safety></li> </ul> | Multiple units | <safety laboratory="" parameter=""> refers safety laboratory parameter for haema biochemistry and coagulation parameter listed in table 18 of the protocol versi. Week 56 cut-off is when all patients for 2-4 have completed visit 13a assessming permanently discontinued treatment. Concizumab (arm 1) data available up week 56 cut-off will be presented.</safety> | atology,<br>ters as<br>on 7.<br>From arm<br>ents or | 5.6.3 |

| Statistical Analys<br>Trial ID: NN741 | | UTN: U1111-1225-9670<br>EudraCT No.: 2018-004889-34 | Date:<br>Version: | 21 July 2022 Status: Final<br>2.0 Page: 24 of 26 | |
|---|---|---|---|---|---|
| Assessment | Change in body weight | On demand (arm 1) • From randomisation (week 0) up until start of concizumab treatment (at least 24 weeks) | kg | Week 56 cut-off is when all patients from arm 2-4 have completed visit 13a assessments or permanently discontinued treatment. Concizumab (arm 1) data available up until week 56 cut-off will be presented. | 5.6.3 |
| | | Concizumab (arm 1) • From start of the new concizumab dosing regimen up until week 56 cut-off | | | |
| | | <ul> <li>Concizumab (arms 2-4)</li> <li>From start of the new concizumab dosing regimen (week 0) up until week 56 cut-off</li> </ul> | | | |
| | | From start of treatment (week 0) to every visit where body weight is planned to be measured up until V13a (week 56) | | | |
| Assessment | Change in systolic blood pressure | On demand (arm 1) • From randomisation (week 0) up until start | mmHg | Week 56 cut-off is when all patients from arm 2-4 have completed visit 13a assessments or permanently discontinued treatment. | 5.6.3 |
| Assessment | Change in diastolic blood pressure | of concizumab<br>treatment (at least 24<br>weeks) | mmHg | Concizumab (arm 1) data available up until week 56 cut-off will be presented. | 5.6.3 |
| Assessment | Change in pulse rate | Concizumab (arm 1) | beats/min | | 5.6.3 |

| Statistical Analys<br>Trial ID: NN741 | | UTN: U1111-1225-9670<br>EudraCT No.: 2018-004889-34 | Date:<br>Version: | 21 July 2022<br>2.0 | | Final<br>of 26 | Novo Nordisk |
|---|---|---|---|---|---|---|---|
| | | From start of the new concizumab dosing regimen up until week 56 cut-off | | | | | |
| | | <ul> <li>Concizumab (arms 2-4)</li> <li>From start of the new concizumab dosing regimen (week 0) up until week 56 cut-off</li> </ul> | | | | | |
| | | From start of treatment (week 0) to every visit where the vital signs are planned to be measured up until V13a (week 56) | | | | | |
| Assessment | Change in physical examination | <ul> <li>Concizumab (arm 1)</li> <li>From start of the new concizumab dosing regimen up until week 56 cut-off</li> <li>Concizumab (arms 2-4)</li> <li>From start of the new concizumab dosing</li> </ul> | % | 2-4 have complete permanently disco | s when all patients from an ed visit 13a assessments or ontinued treatment. 1) data available up until vill be presented. | r | 5.6.3 |
| | | regimen (week 0) up<br>until week 56 cut-off From start of treatment<br>(week 0) to every visit<br>where physical<br>examination is planned to | | | | | |

| Statistical Analysis Plan W56<br>Trial ID: NN7415-4311 | UTN: U1111-1225-9670<br>EudraCT No.: 2018-004889-34 | Date:<br>Version: | 21 July 2022<br>2.0 | Status:<br>Page: | Final 26 of 26 | Novo Nordisk |
|---|---|---|---|---|---|---|
| | be measured up until V13a (week 56) | | | | | |